CLINICAL TRIAL: NCT02451436
Title: Pilot Study of a Sleep and Media Intervention to Improve Adolescents' Metabolic Health and Weight Status
Brief Title: A Sleep and Media Use Intervention to Improve Adolescents' Weight and Risk of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Aaron Fobian, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F150924004
Record Dates: First submitted 2014-12-09; First posted 2015-05-22 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Sleep
Keywords: Adolescents, sleep, media use, obesity, type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep and Media Use Intervention (Active Comparator): The sleep intervention group will receive four sessions including cognitive behavioral training aimed at increasing sleep duration, education on the effects of media use on sleep and problem solving with the participant and parent about increasing sleep duration and decreasing nighttime media use.
  Interventions: Behavioral: Sleep and Media Use Intervention
- Study Skills Control Group (Active Comparator): The control group will receive four sessions of study skills training.
  Interventions: Behavioral: Study Skills Control Group

INTERVENTIONS:
Behavioral: Sleep and Media Use Intervention
  Arms: Sleep and Media Use Intervention
Behavioral: Study Skills Control Group
  Arms: Study Skills Control Group

SUMMARY:
This study aims to assess the effects of a sleep and media intervention on adolescents' overall health.

DETAILED DESCRIPTION:
Introduction. Over the last 30 years, the obesity rate in adolescents has more than tripled, and more than one-third of adolescents were obese in 2010. Many of the complications associated with obesity, including glucose intolerance, hypertension, dyslipidemia and markers of inflammation such as interleukin-6 (IL-6) and C-reactive protein (CRP), are already present in adolescence. The incidence of type 2 diabetes in adolescents has also increased, especially in minorities. Current lifestyle interventions for obesity and type 2 diabetes focused on altering energy balance have not shown promising long-term outcomes. Further research is needed to better understand factors that alter metabolism in order to create more effective interventions.

As obesity and type 2 diabetes rates have risen, adolescents' sleep duration has decreased. Despite requiring more sleep than other children, adolescents often do not obtain adequate sleep. There are many reasons for this decrease in sleep, including delayed circadian rhythm, increased academic demands and extracurricular activities, minimal parental supervision and increased media use. Media use among adolescents has increased significantly over the last 5 years and has been shown to affect adolescents' sleep. It has also been found to be an etiological factor in adolescent obesity.

Experimental studies with adolescents and adults suggest that inadequate sleep duration and poor sleep quality are associated with insulin resistance, glucose intolerance, increased ghrelin and increased markers of inflammation. However, no previous study has successfully examined the effects of a longer-term sleep intervention on factors related to obesity and type 2 diabetes. We propose that short sleep and poor sleep quality may lead to obesity and type 2 diabetes through 2 mechanisms: 1) increased ghrelin, which can lead to increased food intake, decreased energy expenditure and impaired glycemic control, and 2) decreased insulin sensitivity, which also increases insulin. These changes in energy balance and metabolism could lead to weight gain over time and increase adolescents' risk for type 2 diabetes.

Methods. This study aims to assess the effects of a sleep and media use intervention on adolescent body composition, ghrelin and insulin sensitivity. In a randomized controlled trial, 15-17 year olds who are obese and who do not obtain adequate sleep will be randomized to one of two groups: a sleep intervention group or a study skills control group. The sleep intervention group will receive four sessions including cognitive behavioral training aimed at increasing sleep duration, education on the effects of media use on sleep and problem solving with the participant and parent about increasing sleep duration and decreasing nighttime media use. The control group will receive four sessions of study skills training. Sleep duration will be measured by actigraphy, television use will be measured by the TV Allowance device (Family Safe Media, Salt Lake City, UT), and cell phone use will be measured by cellular provider reports and the Break Free mobile application (Mobifolio). Blood draws will be performed 7 days before and after the intervention and at the 3-month follow-up. Body composition will be assessed by dual-energy X-ray absorptiometry (DXA).

Hypotheses and Specific Aims. Primary Aim. Conduct a two-arm parallel group randomized controlled trial of the relative effects of an intervention for adolescent sleep duration and media use on adolescents' sleep duration and quality, insulin sensitivity, appetite-regulating hormones and body composition.

Seven days after the end of the intervention and at the 3-month follow-up, adolescents in the sleep intervention group compared to the control group will have:

H1: Increased sleep duration and sleep quality H2: Increased insulin sensitivity H3: Decreased ghrelin H4: Decreased percent body fat H5: Associations between sleep duration and quality and insulin sensitivity, ghrelin and percent body fat Secondary Aim. Evaluate whether the sleep intervention affects adolescents' nighttime media use.

H1: Adolescents in the sleep intervention group will have decreased nighttime media use (cell phone, internet and television) compared with the control group at both the end of the study and the 3-month follow-up.

Secondary Aim. Evaluate the effects of an intervention for adolescent sleep duration and media use on adolescents' hs-CRP.

Future. Results of this preliminary study will shed light on the impact of a sleep and media use intervention for adolescents in reducing obesity and risk for type 2 diabetes in adolescents. These data will provide support for a future R01 submission testing the effectiveness of a sleep intervention in the context of a larger, well-powered study. It will also provide the foundation for further testing of the mechanisms of action in the relationship between sleep and obesity and type 2 diabetes.

In order to assess the impact of COVID-19 shutdown and virtual school on health, participants who had previously completed at least one blood draw and DXA prior to March 2020 were recruited to complete an additional fasting blood draw and DXA scan in Fall of 2020.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 15-17
* BMI ≥85th percentile
* Android cell phone
* Average normal sleep duration ≤ 7.5 hours

Exclusion Criteria:

* Sleep disorders
* Severe intellectual disability
* Severe mental illness

For the COVID-19 assessment, participants enrolled prior to COVID-19 were eligible for the COVID-19 follow-up visit.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2015-03; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Body composition | Change from baseline body composition to 3 months after intervention and during COVID-19 pandemic if they were enrolled prior to COVID-19
  Assessed through DXA
Ghrelin | Change from baseline to 1 week after the intervention and 3 months after the intervention and during COVID-19 pandemic if they were enrolled prior to COVID-19
  Assessed through blood draw
Insulin | Change from baseline to 1 week after the intervention and 3 months after the intervention and during COVID-19 pandemic if they were enrolled prior to COVID-19
  Assessed through blood draw
Sleep Duration | Change from baseline to 1 week after the intervention and 3 months after the intervention and during COVID-19 pandemic if they were enrolled prior to COVID-19
  Assessed via Actigraphy

SECONDARY OUTCOMES:
Cell Phone Application Use | Change from baseline to 1 week after the intervention and 3 months after the intervention and during COVID-19 pandemic if they were enrolled prior to COVID-19
  Duration of app use
hs-CRP | Change from baseline to 1 week after the intervention and 3 months after the intervention and during COVID-19 pandemic if they were enrolled prior to COVID-19
  Measured via blood draw

CONTACTS AND LOCATIONS:
Locations (1):
- Sparks Center Office of Psychiatric Research, Birmingham, Alabama, United States